CLINICAL TRIAL: NCT07006389
Title: Factors Affecting Response to Extracorporeal Shock Wave Therapy in Plantar Fasciitis: A Cross-sectional Clinical Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Selda Çiftci, Medical Doctor, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 12.31.2024/approval no:4684
Record Dates: First submitted 2025-05-27; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Plantar Fasciitis; Plantar Heel Pain
Keywords: pain; plantar fasciitis; plantar heel pain; ESWT; extracorporeal shock wave therapy
MeSH Terms: conditions — Fasciitis, Plantar; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-responder group to ESWT: Patients who had less than 50% response in the Visual Analog Scale (VAS) after ESWT and patients who had >50% VAS regression in the first month after ESWT and whose pain recurred afterwards
- Responder group to ESWT: Patients who had >50% VAS regression in the 6th month were included in the group that responded to ESWT treatment.

SUMMARY:
Heel pain is a problem that affects daily life activities and quality of life. Extracorporeal shock wave therapy (ESWT) is a treatment used for heel pain. However, some people do not benefit from ESWT treatment. The aim of this study is to determine the factors that affect the response to ESWT in the treatment of heel pain.

DETAILED DESCRIPTION:
Plantar heel pain is one of the reasons that affect daily life activities. There are many treatment methods for this. Extracorporeal shock wave therapy (ESWT) is one of them. However, some patients do not respond to ESWT treatment. In this study, patients were divided into 2 groups as those who did not respond to ESWT treatment in terms of pain (less than 50% decrease in pain level) or those with recurrence of pain and those who responded to treatment. Patients who had passed 3-6 months after ESWT constituted the study groups. These two groups will be compared in terms of age, gender, occupation, weight, height, Body Mass Index (BMI), side: right / left / bilateral, calcaneal angle, Meary angle, presence of spur on X-ray (size in mm if present), dorsiflexion angle degree, plantar fascia thickness with ultrasonography, tibial / plantar nerve conduction study evaluated with electroneuromyography, Visual Analog Scale, Heel Sensitivity Index and Foot Function Index.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Unresponsive to conservative treatments (physical therapy, rest, exercises, anti-inflammatory medical treatment, insoles, etc.)
* Patients who have received ESWT treatment and 3-6 months have passed since ESWT

Exclusion Criteria:

* History of injection therapy including steroids after ESWT treatment
* Those taking NSAIDs in the last 2 weeks
* Those with a history of trauma or surgery to the foot or ankle
* Presence of rheumatic disease affecting the foot or ankle (e.g. spondyloarthritis, etc.)
* Malignancy
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a history of plantar fasciitis
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Calcaneal inclination angle | Day 1
  This angle is established on a weight-bearing lateral foot radiograph between the calcaneal inclination axis (i.e., the lowest portion of the calcaneus) and the supporting horizontal surface. A cut-off point of ≤19° is used to diagnose symptomatic pes planus/flatfoot.
Ankle dorsiflexion degree | Day 1
  The patient is in a prone position with the ankle on the test side away from the base and the leg extended. The therapist will stabilize the tibia. The normal range of ankle dorsiflexion is 20 degrees. Normal plantar flexion is 50 degrees.
Plantar fascia thickness | Day 1
  To be measured by ultrasound; typically shows increased fascial thickness (>4.0 mm) and a hypoechoic fascia.
Tibial/plantar nerve conduction study with electroneuromyography | Day 1
  Nerve conductions show decreased amplitude of the compound muscle action potential (CMAP) of the tibial nerve stimulated at the ankle and recorded from the abductor hallucis and abductor digiti minimi. Sensory and mixed conduction studies are usually performed with centering techniques.

SECONDARY OUTCOMES:
Meary angle | Day 1
  The Meary angle has been used to determine the apex of the deformity on lateral weight-bearing foot radiographs in patients with pes cavus and pes planus. It is the angle between a line drawn through the longitudinal axes of the talus (mid-talus axis) and the first metatarsal (first metatarsal axis). It can be used to classify the severity of the deformity; mild: <15º, moderate: 15-30º, severe: >30º
Plantar calcaneal spurs | Day 1
  Classically, on plain radiography, the presence of a bony spur extending inferomedially from the calcaneus in the sagittal image will be determined, and its size in mm will be determined.
Heel Tenderness index | Day 1
  0=no pain; 1=painful; 2=painful and whines; 3=painful, whines, and withdraws
Foot Function Index | Day 1
  The FFI consists of 23 items divided into 3 subscales that quantify the impact of foot pathology on pain, disability, and activity limitation in patients. Pain, disability, and activity limitation subscale scores range from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Banu Kuran, Professor, MD, Study Director — Şişli Hamidiye Etfal Taining and Research Hospital
Locations (1):
- Şişli Hamidiye Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided